CLINICAL TRIAL: NCT06341192
Title: Clinical Comparison and Motion Analysis of Sports Function Between Combined Anterolateral Ligament Reconstruction With Single Bundle and Double Bundle Anterior Cruciate Ligament Reconstruction
Brief Title: Comparison Between Combined ALLR With Single Bundle and Double Bundle Anterior Cruciate Ligament Reconstruction
Acronym: ALLR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChangGungMH ALL SB DB
Record Dates: First submitted 2024-03-18; First posted 2024-04-02 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-01

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Reconstruction
Keywords: anterior cruciate ligament; anterolateral ligament; single bundle; double bundle; optical motion capture; graft rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Single-Bundle ACL + ALL Reconstruction Group:
  * Patients in this group will undergo reconstruction of the anterior cruciate ligament (ACL) using a single-bundle graft technique.
  * In addition, they will have the anterolateral ligament (ALL) reconstructed using a portion of the same graft material.
  * For the ALL reconstruction, a commonly used technique is the Sonnery-Cottet ALL reconstruction using a split graft.
  Double-Bundle ACL + ALL Reconstruction Group:
  * Patients in this group will undergo anatomic double-bundle ACL reconstruction using two graft bundles to more anatomically replicate the native ACL's anteromedial and posterolateral bundles.
  * Like the single-bundle group, they will also have supplemental ALL reconstruction performed using a portion of the graft material.
  * The double-bundle ACL reconstruction aims to better restore the ACL's complex anatomic footprint and bundles' tension patterns.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Double bundle ACL combined anterolateral ligament reconstruction (Experimental): ACL reconstruction with triple folded semitendinosus and non folded gracilis and fibertape
  Interventions: Procedure: Double-bundle ACL combined anterolateral ligament reconstruction
- Single bundle ACL combined anterolateral ligament reconstruction (Experimental): Single bundle ACL combined anterolateral ligament reconstruction
  Interventions: Procedure: Single-bundle ACL combined anterolateral ligament reconstruction

INTERVENTIONS:
Procedure: Single-bundle ACL combined anterolateral ligament reconstruction — Single-Bundle ACL + ALL Reconstruction Group:
  Patients in this group will undergo reconstruction of the anterior cruciate ligament (ACL) using a single-bundle graft technique.
  In addition, they will have the anterolateral ligament (ALL) reconstructed using a portion of the same graft material.
  The single ACL bundle is typically positioned to replicate the anatomic footprint of the native ACL.
  For the ALL reconstruction, a commonly used technique is the Sonnery-Cottet ALL reconstruction using a gracilis tendon graft.
  This combines an intra-articular ACL reconstruction with an extra-articular lateral tenodesis to improve rotational instability.
  Arms: Single bundle ACL combined anterolateral ligament reconstruction
Procedure: Double-bundle ACL combined anterolateral ligament reconstruction — Double-Bundle ACL + ALL Reconstruction Group:
  Patients in this group will undergo anatomic double-bundle ACL reconstruction using two graft bundles to more anatomically replicate the native ACL's anteromedial and posterolateral bundles.
  Like the single-bundle group, they will also have supplemental ALL reconstruction performed using a portion of the graft material.
  The double-bundle ACL reconstruction aims to better restore the ACL's complex anatomic footprint and bundles' tension patterns.
  Arms: Double bundle ACL combined anterolateral ligament reconstruction

SUMMARY:
The goal of this clinical trial is to test and compare different surgical techniques in patients with anterior cruciate ligament (ACL) injuries. The main questions it aims to answer are:

* What are the optimal criteria for selecting between single-bundle ACL reconstruction combined with anterolateral ligament (ALL) reconstruction versus double-bundle ACL reconstruction combined with ALL reconstruction?
* How do these two surgical techniques compare in terms of post-operative knee stability, functional outcomes, and reducing re-tear rates?

Participants will:

* Undergo pre-operative MRI imaging, ligament stability testing, and motion analysis evaluations
* Be randomly assigned to either:

  * Single-bundle ACL + ALL reconstruction
  * Double-bundle ACL + ALL reconstruction
* Receive the assigned surgical procedure
* Participate in post-operative follow-ups, ligament stability testing, and motion analysis at 6 months and 1 year

Researchers will compare the single-bundle ACL + ALL group and the double-bundle ACL + ALL group to see if one technique demonstrates superior knee stability, functional outcomes (e.g. return to sport ability), and lower ACL re-tear rates.

DETAILED DESCRIPTION:
Anterolateral ligament(ALL) combined with anterior cruciate ligament reconstruction(ACL) has become more and more popular in recent years, as ALL could protect the ACL graft in tibial internal rotation, and prevent the ACL graft from rupture. Cottet et al. proposed a minimal invasive method with Y-figure construct of ALL, without acquiring additional graft from the patient. Their data showed significant lower graft re-rupture rate and faster return-to-sport(RTS). There are many different techniques of ACL combined ALL reconstruction. While these methods mostly are single bundle ACL combined ALL reconstruction. Previous cadaver studies told that the anterior cruciate ligament is composed of anteromedial and posterolateral bundle. It had been debated between single bundle and double bundle ACL reconstruction for years. As a result, it is meaningful to compare the clinical outcomes between ALL combined with single bundle or double bundle ACL reconstruction. Our studies included MRI image, arthrometer measurement and optical motion capture system. We hope to compare the clinical outcomes and sports function between A: single bundle ACL combined ALL reconstruction and B: double bundle ACL combined ALL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients plan to receive ACL surgery
* at least 18 years old

Exclusion Criteria:

* Presented history of the injured leg or congenital abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Patient-reported outcome measures (PROMs) | Preoperative, 3 months, 6 months, 9 months, 1 year
  International Knee Documentation Committee (IKDC) subjective score. The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Patient-reported outcome measures (PROMs) | Preoperative, 3 months, 6 months, 9 months, 1 year
  Marx's activity score;The Marx Scale consists of four questions concerning four activities or actions: running, cutting, deceleration, and pivoting. The patient or survey respondent is asked to report on the frequency with which they performed the activity in their healthiest state within the past year. From 0 point(the worst) to 16 points(the best).
Patient-reported outcome measures (PROMs) | Preoperative, 3 months, 6 months, 9 months, 1 year
  SANE score, The Single Assessment Numeric Evaluation (SANE) is a patient rating from 0-100. Patients rate their current illness score in relation to their pre-injury baseline
Knee ligament stability: | Preoperative, 6 months, 1 year
  Anterior tibial translation measured using a ligament arthrometer (GNRB) to objectively quantify anteroposterior knee laxity
Knee ligament stability clinical evaluation | Preoperative, 6 months, 1 year
  Lachman test
Knee ligament stability clinical evaluation | Preoperative, 6 months, 1 year
  pivot shift test
Knee ligament stability clinical evaluation | Preoperative, 6 months, 1 year
  Anterior drawer test
Functional performance and return to sport | Preoperative, 6 months, 1 year
  Lower limb muscle strength
Functional performance and return to sport | Preoperative, 6 months, 1 year
  Lower limb symmetry index
Imaging | Preoperative, 1 year
  Pre- and post-operative X-ray analysis to assess bone tunnels position
Imaging | Preoperative, 1 year
  Pre- and post-operative MRI analysis to assess graft ligamentization.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Pang Dr. Yang, Principal Investigator — Cheng Gung memorial hospital
Locations (1):
- Chang Gung memorial hospital, Taoyuan District, taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No
1. Protection of participant privacy and confidentiality is paramount in this study involving sensitive medical data and procedures. Sharing identifiable IPD could breach the trust and privacy of these patients undergoing knee surgeries.
  2. The informed consent process likely did not explicitly state or obtain approval from participants to share their individual-level data, including medical images, functional assessments, and clinical outcomes, with third parties outside the research team.

REFERENCES:
- [Background] Cameron KL, Peck KY, Davi SM, Owens CRBD, Svoboda CRSJ, DiStefano LJ, Marshall SW, de la Motte SJ, Beutler CRAI, Padua DA. Association Between Landing Error Scoring System (LESS) Items and the Incidence Rate of Lower Extremity Stress Fracture. Orthop J Sports Med. 2022 Jun 9;10(6):23259671221100790. doi: 10.1177/23259671221100790. eCollection 2022 Jun. PMID 35706554
- [Background] Helito CP, Helito PVP, Costa HP, Demange MK, Bordalo-Rodrigues M. Assessment of the Anterolateral Ligament of the Knee by Magnetic Resonance Imaging in Acute Injuries of the Anterior Cruciate Ligament. Arthroscopy. 2017 Jan;33(1):140-146. doi: 10.1016/j.arthro.2016.05.009. Epub 2016 Jun 17. PMID 27324971
- [Background] Sonnery-Cottet B, Thaunat M, Freychet B, Pupim BH, Murphy CG, Claes S. Outcome of a Combined Anterior Cruciate Ligament and Anterolateral Ligament Reconstruction Technique With a Minimum 2-Year Follow-up. Am J Sports Med. 2015 Jul;43(7):1598-605. doi: 10.1177/0363546515571571. Epub 2015 Mar 4. PMID 25740835
- [Background] Batty LM, Firth A, Moatshe G, Bryant DM, Heard M, McCormack RG, Rezansoff A, Peterson DC, Bardana D, MacDonald PB, Verdonk PCM, Spalding T, Getgood AMJ; STABILITY Study Group; Willits K, Birmingham T, Hewison C, Wanlin S, Firth A, Pinto R, Martindale A, O'Neill L, Jennings M, Daniluk M, Boyer D, Zomar M, Moon K, Pritchett R, Payne K, Fan B, Mohan B, Buchko GM, Hiemstra LA, Kerslake S, Tynedal J, Stranges G, Mcrae S, Gullett L, Brown H, Legary A, Longo A, Christian M, Ferguson C, Mohtadi N, Barber R, Chan D, Campbell C, Garven A, Pulsifer K, Mayer M, Simunovic N, Duong A, Robinson D, Levy D, Skelly M, Shanmugaraj A, Howells F, Tough M, Thompson P, Metcalfe A, Asplin L, Dube A, Clarkson L, Brown J, Bolsover A, Bradshaw C, Belgrove L, Millan F, Turner S, Verdugo S, Lowe J, Dunne D, McGowan K, Suddens CM, Declercq G, Vuylsteke K, Van Haver M. Association of Ligamentous Laxity, Male Sex, Chronicity, Meniscal Injury, and Posterior Tibial Slope With a High-Grade Preoperative Pivot Shift: A Post Hoc Analysis of the STABILITY Study. Orthop J Sports Med. 2021 Apr 6;9(4):23259671211000038. doi: 10.1177/23259671211000038. eCollection 2021 Apr. PMID 33889648
- [Background] Sonnery-Cottet B, Daggett M, Fayard JM, Ferretti A, Helito CP, Lind M, Monaco E, de Padua VBC, Thaunat M, Wilson A, Zaffagnini S, Zijl J, Claes S. Anterolateral Ligament Expert Group consensus paper on the management of internal rotation and instability of the anterior cruciate ligament - deficient knee. J Orthop Traumatol. 2017 Jun;18(2):91-106. doi: 10.1007/s10195-017-0449-8. PMID 28220268